CLINICAL TRIAL: NCT04529408
Title: EARSATS-19: In-ear Measurement of Blood Oxygen Saturation in COVID-19 Follow up
Acronym: EARSATS-19
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 285603
Record Dates: First submitted 2020-08-26; First posted 2020-08-27 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Covid19; Pulmonary Disease
MeSH Terms: conditions — COVID-19; Lung Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 Follow up clinic: Patients attending routine post-COVID-19 follow up clinic
  Interventions: Device: EarSats Pulse Oximeter Probe
- Pulmonary Disease clinic: Patients attending routine outpatient appointment for pulmonary disease
  Interventions: Device: EarSats Pulse Oximeter Probe

INTERVENTIONS:
Device: EarSats Pulse Oximeter Probe — Off-the-shelf pulse oximeter embedded into a memory foam ear plug for measuring blood oxygen saturation (SpO2) from the ear canal; in-ear SpO2 measured at-rest and during 6 minute walk test

SUMMARY:
TITLE EARSATS-19: In-ear measurement of blood oxygen saturation in COVID-19 follow up

DESIGN Non-inferiority study

AIMS To evaluate qualitative and quantitative performance of in-ear SpO2 monitoring against the gold standard right finger-clip pulse oximeter -- towards validation for use in COVID-19 in the acute ambulatory and long-term monitoring setting

OUTCOME MEASURES

In-ear SpO2 compared with gold-standard finger-clip pulse oximeter:

Correlation between SpO2 measurements at rest Correlation between SpO2 measurements during 6 minute walk test Signal quality during 6 minute walk test Qualitative evaluation of clinical and patient user acceptability using questionnaires

POPULATION 30 patients attending COVID-19 follow-up clinic and 30 patients with chronic lung disease attending routine outpatient investigations

ELIGIBILITY Aged 18 and above, no upper age limit Able to give informed consent No abnormal ear anatomy.

DURATION 12 months

DETAILED DESCRIPTION:
Non-invasive ambulatory estimation of blood oxygen saturation (SpO2) has emerged as an important clinical requirement to detect hypoxia (low blood oxygen) in the delayed post-infective phase of COVID- 19, where dangerous hypoxia may occur in the absence of subjective breathlessness. This now commonly termed 'silent' hypoxia presents an immediate clinical driver.

The COVID-19 pandemic places substantial pressure on clinical resources with ambulatory patients who were often discharged home to be cared for on virtual wards with daily telephone consults. Now the initial surge has settled, we are beginning to understand the challenge of following up patients who have had COVID-19 at volumes that mean doing this in a timely fashion is not possible (BTS Guidance 6 weeks).

There is mounting concern that the huge number of COVID-19 survivors will be at increased risk of chronic lung diseases such as pulmonary fibrosis, where early capture of patterns of low SpO2 could unearth desperately needed insights for preventing disease progression. The inconveniences, impracticalities and inaccuracies of conventional measurement of SpO2 (the percentage unit of blood oxygen) using a conventional finger probe for discrete readings are well established. A user-friendly, remote continuous SpO2 monitoring tool would therefore allow the rapid identification of any deterioration post discharge and also track longer-term recovery, allowing the accurate triage of patients to limited follow up resources.

Hearables and In-Ear Photoplethysmography

Reflective photoplethysmography (PPG), which uses a changes in the ratio between red and infrared light to estimate SpO2, can be measured from any site with skin that has vasculature, but for SpO2 measurement has conventionally been from fingers or sometimes the earlobe. The recent interest in the development of Hearables9 has promoted the ear canal as a preferred site for the measurement of vital signs in digital health technology. Indeed, the ear canal, which acts as a shield from external electrical noise (resembling a nature-built Faraday cage), represents a unique opportunity for physiological measurements, due to its general fixed position relative to the heart (ear-electrocardiogram) and proximity to the brain (ear-electroencephalogram). Relative to limbs, the head moves less in daily life and this is one property that has helped establish the feasibility of wearables to detect Ear-ECG and Ear-EEG.

Unlike the finger and ear lobe PPG signal, in-ear PPG has shown that the ear canal, owing to being a narrow cavity with consistent blood supply, offers a signal which is stable and resistant to changes in blood volume occurring during hypothermia . This attribute has established the ear canal as a preferred site for accurate core body temperature measurement. In-ear PPG has also been shown to be far more sensitive than earlobe and finger PPG to amplitude variations that arise from respiration, thus allowing for a better measurement of respiratory rate. Furthermore, a significant delay has been evidenced between earlobe pulse oximetry and pulse oximetry on the hand or the foot for detection of hypoxemia (low levels of blood oxygen)..

Previous work led by Professor Mandic's group in the Faculty of Engineering showed that in a study of 14 healthy volunteers in-ear PPG compared with the current standard of care - the finger clip -- the in-ear sensor shows non-inferiority and potential superiority with regard to detection of a mean blood oxygen delay (the time it took from detecting minimal blood oxygen change in the ear to detecting minimal blood oxygen in the finger) reduction of 12.4 seconds, thus being faster at identifying acute desaturation.

RATIONALE FOR CURRENT STUDY

This project sets out to establish the feasibility of SpO2 measurement from the ear canal as a convenient site for monitoring in the post COVID-19 follow up patient population, and perform a comprehensive comparison with the right index finger - the conventional clinical measurement site. The initial phase of the study will start with a total of n = 60 patients; 30 patients, who will be attending hospital as part of their routine clinical post COVID-19 follow up, which already includes SpO2 monitoring and a six minute walk test (6MWT). This study will also recruit a further 30 patients with chronic lung disease also attending for these routine outpatient investigations.

The continuous monitoring and rapid detection of desaturation can provide earlier warning of deterioration or detailed tracking of an improving trajectory. Current alternative monitoring strategies are reactive and all revolve around the classical finger or earlobe clip, which are less sensitive and present a number of challenges for continual monitoring. Living daily life with a finger clip, or even an earlobe clip, is problematic with much higher signal noise from movement artefacts with the finger clip compared to the ear bud placed within a stable head position.

From a patient perspective, the ear bud form factor that will be used in this study is familiar to them, being similar to an in-ear headphone, and will be much less intrusive to daily activities than a finger clip. Therefore the potential for continuous monitoring during the active day and the night time is much more user-friendly, and vital for the younger and potentially more active COVID-19 patients. Continuous monitoring would allow the development of protocolised management pathways to provide increasing levels of supported self-care to patients, freeing up vital resources during future pandemics.

The data generated in this pilot feasibility study would allow scaling to prepare for larger research projects in any subsequent surge discharge and follow up. The next stage would move to outpatient monitoring, with ambulatory patients going home with the device and the incorporation of further COVID patient populations such as inpatients being monitored for deterioration, where these devices could provide accurate continuous monitoring of SpO2, detecting any deterioration before they develop breathlessness and their condition becomes life threatening. This project therefore directly complements the NHS' strategic priority for early supported discharge monitoring for COVID-19 positive patients and follow up for long-term complications.

The COVID-19 follow up clinic cohort (n = 30) is ideally placed to evaluate this technology; from a quantitative point of view, a significant number of these patients will likely experience desaturation during the 6MWT, serving as an opportunity to test the device's ability to detect this. Qualitatively, since many of these patients will have either had hospital admissions or home monitoring -- and therefore lived experience of SpO2 monitoring -- they are uniquely qualified to offer valuable input on user experience. Similarly, the chronic lung disease cohort (n = 30), attending for routine OP baseline SpO2 measurement and 6MWT are also well-suited to this study.

In the long term this technology will also prove an invaluable device for the home monitoring of respiratory patients. Beyond the current pandemic there exists a general quest for more personalised health data, such that pulse oximetry measurement of capillary oxygen saturation (SpO2) will likely expand into both the clinical and consumer market of wearable health technology in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending respiratory clinic either for COVID-19 follow up or for chronic lung disease.
* Able to give informed consent (where not able to use CIE, paper consent form will be made available)

Exclusion Criteria:

* Abnormal ear canal anatomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatient population attending either COVID-19 follow up or chronic respiratory disease clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-08-26 (Actual); Primary Completion 2022-08-10 (Actual); Study Completion 2022-08-10 (Actual)

PRIMARY OUTCOMES:
In-Ear vs finger SpO2 | 12 months for full participant recruitment (actual head-to head comparison takes 1 minute for baseline reading and 6 minutes for 6-min walk test per patient)
  Mean error and root mean square error; measurements for statistical significance using a paired t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Peters, MD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College Healthcare NHS Trust, London, Non-US/Non-Canadian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Held within Imperial College London as per standard local data protection guidelines. Data may be considered for sharing upon reasonable request.

REFERENCES:
- [Background] Goverdovsky V, von Rosenberg W, Nakamura T, Looney D, Sharp DJ, Papavassiliou C, Morrell MJ, Mandic DP. Hearables: Multimodal physiological in-ear sensing. Sci Rep. 2017 Jul 31;7(1):6948. doi: 10.1038/s41598-017-06925-2. PMID 28761162